CLINICAL TRIAL: NCT02963064
Title: A Phase 1/2 Study to Evaluate the Safety, Tolerability, and Efficacy of JSP191 for Hematopoietic Cell Transplantation Conditioning to Achieve Engraftment and Immune Reconstitution in Subjects With SCID
Brief Title: JSP191 Antibody Targeting Conditioning in SCID Patients
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor Decision - terminated due to changes in company priorities and not related to safety concerns.
Sponsor: Jasper Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JAS-BMT-CP-001
Record Dates: First submitted 2016-11-02; First posted 2016-11-15 (Estimated); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: SCID
Keywords: Immunodeficiency; Pediatric; SCID; Bone Marrow Transplantation; GVHD; Stem Cells; Chimerism; Transplant; BMT
MeSH Terms: conditions — Immunologic Deficiency Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Blood Stem Cell Transplant w/ anti-CD117 conditioning (Experimental): The study will enroll two groups: Group A: previously transplanted SCID patients; Group B: newly diagnosed SCID. The study plans to assess JSP191 in different dose cohorts. Patients will receive a single dose of intravenous JSP191 antibody followed by monitoring for antibody clearance. Once the antibody has cleared below a certain level, patients will receive stem cell transplant and be monitored for hematopoietic recovery.
  Interventions: Biological: Humanized anti-CD117 Monoclonal Antibody (JSP191)

INTERVENTIONS:
Biological: Humanized anti-CD117 Monoclonal Antibody (JSP191) — Procedure: single intravenous infusion of JSP191 antibody

SUMMARY:
A Phase 1/2 study to evaluate the safety, tolerability, and efficacy of an antibody conditioning regimen, known as JSP191, in patients with Severe Combined Immune Deficiency undergoing blood stem cell transplantation

DETAILED DESCRIPTION:
A Phase 1/2 study to evaluate the safety, tolerability, and efficacy of an antibody conditioning regimen, known as JSP191, in patients with SCID undergoing blood stem cell transplantation. Blood Stem Cell transplantation offers the only potentially curative therapy for SCID.

The biological conditioning regimen, JSP191, is an antibody that binds to CD117. CD117 is the receptor for Stem Cell Factor on blood forming cells. CD117 binding to Stem Cell Factor is critical for survival and maintenance of blood forming stem cells. The binding of JSP191 to CD117 blocks CD117 from binding to Stem Cell Factor on blood forming stem cells. In the absence of CD117/Stem Cell Factor binding, hematopoietic stem cells that are currently occupying the bone marrow niches in SCID patients exit from the bone marrow.

ELIGIBILITY:
Key Inclusion Criteria:

1. Typical SCID as defined by Primary Immune Deficiency Treatment Consortia including but not limited to the following subtypes:

   1. T-, B+, NK-: IL-2Rcγ deficient, JAK3-deficient (no longer enrolling)
   2. T-, B-, NK+: RAG1/2 deficient, Artemis-deficient
   3. T-, B+, NK+: IL7Rα deficient, CD3 subunit deficient, CD45 deficient (no longer enrolling) OR Variant SCID with absent or low T cell function, Omenn syndrome, Leaky SCID, Reticular dysgenesis, Adenosine deaminase deficiency, and Purine nucleoside phosphorylase deficiency may be included after consultation with the medical monitor.
2. Patients with human leukocyte antigen (HLA) matched related or unrelated donors
3. Adequate end organ function as defined in study protocol
4. Age ≤ 12 years
5. Prior donor of appropriate age (≥ 5 years old) available for re-collection of stem cells
6. Previous allogeneic Hematopoietic Cell Transplantation HCT (≥ 6 months post initial transplant) with poor graft function

Key Exclusion Criteria:

1. Patients with any acute or uncontrolled infections
2. Patients receiving any other investigational agents, or concurrent biological, chemotherapy, or radiation therapy
3. Patients with active malignancies
4. Active GVHD within 6 months prior to enrollment, or on immunosuppressive therapy for GVHD

Ages: 3 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2025-07-07 (Actual); Study Completion 2025-07-07 (Actual)

PRIMARY OUTCOMES:
Phase 1: Safety and tolerability of JSP191 as conditioning therapy in SCID patients undergoing HCT: adverse events | Up to 5 years post Donor Cell Transplant (28 days dose limiting toxicity period)
  The number of subjects experiencing dose limiting toxicities including adverse events and serious adverse events will be assessed.
Phase 2: Efficacy of JSP191 as conditioning therapy in SCID patients | Up to 24 weeks post Donor Cell Transplant
  To enable engraftment of allogeneic CD34+ hematopoietic cells, as determined by CD15+ donor myeloid chimerism
Phase 2: Efficacy of JSP191 as conditioning therapy in SCID patients | Weeks 36-104 post Donor Cell Transplant
  To enable immune reconstitution, as determined by the production of naive T cells

CONTACTS AND LOCATIONS:
Overall Officials: Rajni A. Agarwal-Hashmi, M.D., Principal Investigator — Lucile Packard Children's Hospital; Christopher C. Dvorak, M.D., Principal Investigator — UCSF Benioff's Children's Hospital; Joseph H. Oved, M.D., Principal Investigator — Memorial Sloan Kettering Cancer Center; Theodore B. Moore, M.D., Principal Investigator — University of California, Los Angeles; Sharat Chandra, M.D., Principal Investigator — Children's Hospital Medical Center, Cincinnati; Christen L Ebens, M.D., MPH, Principal Investigator — University of Minnesota; Harry L Malech, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC); Shanmuganathan Chandrakasan, M.D., Principal Investigator — Children's Healthcare of Atlanta; Neena Kapoor, M.D., Principal Investigator — Children's Hospital Los Angeles; Elizabeth D Hicks, M.D., Principal Investigator — Children's National Research Institute; Susan Prockop, M.D., Principal Investigator — Boston Children's Hospital
Locations (9):
- United States (9):
  - UCLA Mattel Children's Hospital, Los Angeles, California
  - Lucile Packard Children's Hospital, Palo Alto, California
  - UCSF Benioff's Children's Hospital, San Francisco, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - University of Minnesota, Minneapolis, Minnesota
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No
Data collected is for future publication